CLINICAL TRIAL: NCT06341374
Title: Impact of Sleep Disorders on Innate Immunity in COVID-19 Patients. A Cohort Study
Brief Title: Impact of Sleep Disorders on Innate Immunity in COVID-19 Patients
Status: Recruiting | Type: Observational
Sponsor: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Andrea Grau Freixinet, Pulmonology medical specialist, Parc Taulí Hospital Universitari
Other Study IDs: 2023/5079
Record Dates: First submitted 2024-03-29; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Apnea, Obstructive Sleep; SARS CoV 2 Infection
Keywords: Obstructive Sleep Apnea; Innate immunity; SARS-CoV-2
MeSH Terms: conditions — Sleep Apnea, Obstructive; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants who have had severe COVID-19 infection with sleep disturbance: This cohort of participants will be recruited from participants in ongoing study in our institution (CEIm 2021/5096) where exploring contributions of sleep disorders on severity of COVID-19.
  To explore present sleep status participants will be asked to fill out sleep questionnaires referred to their sleep characteristics since COVID-19 episode until present moment. As objective evaluation of sleep participants will perform a night home sleep study with WatchPAT® 300 sleep recording, Itamar Medical Ltd.
  Cohort 1 will be those participants who have had a severe COVID19 infection and have been diagnosed with a sleep disorder.
  Interventions: Biological: Influvac Tetra
- Participants who have had severe COVID-19 infection without sleep disorder: Participants with severe COVID19 infection and no currently diagnosed sleep disorders
  Interventions: Biological: Influvac Tetra
- Participants who have had mild COVID-19 infection with sleep disturbance: Participants who have had a mild COVID19 infection and have been diagnosed with a sleep disorder
  Interventions: Biological: Influvac Tetra
- Participants who have had mild COVID-19 infection without sleep disorder: Participants who have had a mild COVID19 infection and have not been diagnosed with a sleep disorder
  Interventions: Biological: Influvac Tetra

INTERVENTIONS:
Biological: Influvac Tetra — All participants will take influenza vaccine (Influvac Tetra, Abbott Biologicals, IL, USA) and the trained immune response will be evaluated.

SUMMARY:
Sleep is an important modulator of the immune response, whereby sleep disturbances (ie, poor sleep quality, insufficient sleep and/or primary sleep disorder, obstructive sleep apnea (OSA)) contribute to inflammatory disease risk and dysregulation of immune response in front of infectious agents.

The objective of this study is to evaluate the impact of undiagnosed and non-treated sleep disorders on innate immunity in a cohort of COVID-19 patients and the role of trained immunity induced by influenza vaccination in the innate immune response.

DETAILED DESCRIPTION:
Sleep and immune system have reciprocal relationship. Sleep has a restorative role on immune system, influencing innate and adaptive immunity and sleep disorders can decrease immune response.

Healthy innate immunity is crucial into regulation of the response against SARS-CoV-2.

The hypothesis of the study is that the innate immunity response is blunted by sleep disorders and, this mitigated immune response, could influence on COVID-19 severity. Impaired immune response in patients with sleep disorders could be ameliorated inducing trained immunity by influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years old with diagnosis of COVID-19 during first year of coronavirus pandemic in March-June 2021.

Exclusion Criteria:

* >70 years and <18 years
* Recent COVID-19 (<6 months)
* Other infection (<3 months)
* Obstructive sleep apnea in treatment with CPAP prior to COVID infection.
* Immunosuppressed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the local cohort database COVID-19 (Department of Epidemiology) which includes those patients who received medical care at the Hospital Universitari Parc Taulí during the first year of the coronavirus pandemic in March-June 2021.
  Participants will be classified with or without sleep disorders based on the results of nocturnal pulse oximetry (WatchPAT).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Immunological study: cytokines. | To evaluate immune response blood samples will be taken at the time influenza vaccine is given, 7 and 30 days later.
  To measure in blood: IL-1 beta, IL-6, IL-8, IL-10, TNF-alfa, IFN-alfa, IFN-gamma, GM-CSF.

SECONDARY OUTCOMES:
Innate cells: monocytes, classical dendritic cells and Natural Killer cells. | To evaluate immune response blood samples will be taken at the time influenza vaccine is given, 7 and 30 days later.
  To measure: monocytes (CD45, CD14, CD16, HLA-DR), classical dendritic cells (CD45, CD1c, CD141, CD11c, CD86) and NK cells (CD45, CD56, CD16, Pan-KIR2D, NKG2D
Epigenetic modification. | To evaluate immune response blood samples will be taken at the time influenza vaccine is given, 7 and 30 days later.
  To measure: H3K4me3, H3K4me1 and H3K27Ac
Diagnostic of obstructive sleep apnea in selected cohort | It is an overnight study that will last for one night.
  Night home sleep study with WatchPAT® 300.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose M Masdeu, Medicine, Principal Investigator — Hospital Universitari Parc Tauli, Sabadell; Andrea F Grau, Medicine, Principal Investigator — Hospital Universitari Parc Tauli, Sabadell
Locations (1):
- Hospital Universitari Parc Tauli, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borbely AA, Daan S, Wirz-Justice A, Deboer T. The two-process model of sleep regulation: a reappraisal. J Sleep Res. 2016 Apr;25(2):131-43. doi: 10.1111/jsr.12371. Epub 2016 Jan 14. PMID 26762182
- [Background] Irwin MR, Opp MR. Sleep Health: Reciprocal Regulation of Sleep and Innate Immunity. Neuropsychopharmacology. 2017 Jan;42(1):129-155. doi: 10.1038/npp.2016.148. Epub 2016 Aug 11. PMID 27510422
- [Background] Besedovsky L, Lange T, Haack M. The Sleep-Immune Crosstalk in Health and Disease. Physiol Rev. 2019 Jul 1;99(3):1325-1380. doi: 10.1152/physrev.00010.2018. PMID 30920354
- [Background] Spiegel K, Sheridan JF, Van Cauter E. Effect of sleep deprivation on response to immunization. JAMA. 2002 Sep 25;288(12):1471-2. doi: 10.1001/jama.288.12.1471-a. No abstract available. PMID 12243633
- [Background] Partinen M, Holzinger B, Morin CM, Espie C, Chung F, Penzel T, Benedict C, Bolstad CJ, Cedernaes J, Chan RNY, Dauvilliers Y, De Gennaro L, Han F, Inoue Y, Matsui K, Leger D, Cunha AS, Merikanto I, Mota-Rolim S, Nadorff M, Plazzi G, Schneider J, Sieminski M, Wing YK, Bjorvatn B. Sleep and daytime problems during the COVID-19 pandemic and effects of coronavirus infection, confinement and financial suffering: a multinational survey using a harmonised questionnaire. BMJ Open. 2021 Dec 13;11(12):e050672. doi: 10.1136/bmjopen-2021-050672. PMID 34903540
- [Background] Park SH. An Impaired Inflammatory and Innate Immune Response in COVID-19. Mol Cells. 2021 Jun 30;44(6):384-391. doi: 10.14348/molcells.2021.0068. PMID 34098591
- [Background] Netea MG, Giamarellos-Bourboulis EJ, Dominguez-Andres J, Curtis N, van Crevel R, van de Veerdonk FL, Bonten M. Trained Immunity: a Tool for Reducing Susceptibility to and the Severity of SARS-CoV-2 Infection. Cell. 2020 May 28;181(5):969-977. doi: 10.1016/j.cell.2020.04.042. Epub 2020 May 4. PMID 32437659
- [Background] Netea MG, Quintin J, van der Meer JW. Trained immunity: a memory for innate host defense. Cell Host Microbe. 2011 May 19;9(5):355-61. doi: 10.1016/j.chom.2011.04.006. PMID 21575907
- [Background] Laupeze B, Del Giudice G, Doherty MT, Van der Most R. Vaccination as a preventative measure contributing to immune fitness. NPJ Vaccines. 2021 Jul 27;6(1):93. doi: 10.1038/s41541-021-00354-z. PMID 34315886
- [Background] Wagstaffe HR, Pickering H, Houghton J, Mooney JP, Wolf AS, Prevatt N, Behrens RH, Holland MJ, Riley EM, Goodier MR. Influenza Vaccination Primes Human Myeloid Cell Cytokine Secretion and NK Cell Function. J Immunol. 2019 Sep 15;203(6):1609-1618. doi: 10.4049/jimmunol.1801648. Epub 2019 Aug 19. PMID 31427444
- [Background] Debisarun PA, Gossling KL, Bulut O, Kilic G, Zoodsma M, Liu Z, Oldenburg M, Ruchel N, Zhang B, Xu CJ, Struycken P, Koeken VACM, Dominguez-Andres J, Moorlag SJCFM, Taks E, Ostermann PN, Muller L, Schaal H, Adams O, Borkhardt A, Ten Oever J, van Crevel R, Li Y, Netea MG. Induction of trained immunity by influenza vaccination - impact on COVID-19. PLoS Pathog. 2021 Oct 25;17(10):e1009928. doi: 10.1371/journal.ppat.1009928. eCollection 2021 Oct. PMID 34695164